CLINICAL TRIAL: NCT01655862
Title: Multi-Centre, Prospective, Observational Study of Patient Reported Outcomes in Patients Diagnosed With Cervical Dystonia and Treated With OnabotulinumtoxinA for Injection (BOTOX®) (POSTURe)
Brief Title: A Prospective, Observational Study of Patients With Cervical Dystonia (Dystonie) Treated With OnabotulinumtoxinA
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: CMA-BTX-12-001
Record Dates: First submitted 2012-07-31; First posted 2012-08-02 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Torticollis
MeSH Terms: conditions — Torticollis | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- OnabotulinumtoxinA: OnabotulinumtoxinA injections at doses and frequencies as determined by the physician in accordance with clinical practice.
  Interventions: Biological: OnabotulinumtoxinA

INTERVENTIONS:
Biological: OnabotulinumtoxinA — OnabotulinumtoxinA injections at doses and frequencies as determined by the physician in accordance with clinical practice.
  Other Names: botulinum toxin Type A; BOTOX®

SUMMARY:
This is an observational study to assess health-related quality of life in patients with cervical dystonia (dystonie) treated with OnabotulinumtoxinA per routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cervical dystonia (dystonie) and able to receive botulinum toxin Type A as deemed medically necessary by the physician

Exclusion Criteria:

* Participation in a clinical trial for any botulinum toxin indication
* Planning elective surgery during the observational study period
* Treatment with any botulinum toxin product for cervical dystonia (dystonie)
* Treatment with any botulinum toxin product for a non-cervical dystonia (dystonie) condition within 2 months of study start

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Cervical Dystonia (Dystonie)
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2012-07; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Cervical Dystonia Impact Profile Questionnaire (CDIP-58) Score | Baseline, 96 Weeks

SECONDARY OUTCOMES:
Patient's Global Impression of Change (PGIC) Using a 7-Point Scale | Baseline, 96 Weeks
Work Productivity Assessment Using a 10-Item Questionnaire | 96 Weeks
Change from Baseline in Hospital Anxiety and Depression Scale (HAD) Score | Baseline, 96 Weeks
Reasons for Withdrawal of Treatment | 96 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Goran Davidovic, Study Director — Allergan
Locations (8):
- Canada (8):
  - Clinique Neuro-Rive Sud, Greenfield Park, Quebec
  - Hôpital Maisonneuve-Rosemont, Montreal, Quebec
  - Chum-Notre-Dame, Montreal, Quebec
  - Queen Elizabeth Health Centre: Medical Specialist Clinic, Montreal, Quebec
  - CHU de Québec, Hôpital de l'Enfant-Jésus, Québec, Quebec
  - Centre Medical Le Mesnil, Québec, Quebec
  - Polyclinique Medicale des Ponts, Saint Romuald, Quebec
  - CHU - Sherbrooke, Sherbrooke, Quebec